CLINICAL TRIAL: NCT05208658
Title: Evaluate Objectively the Change in the Vergence Responses of Binocular and Accommodative Normal Subjects After Performing a Classic Vision Therapy Protocol
Brief Title: Characteristics of the Vergence Responses of Binocularly Normal Subjects After a Vision Therapy Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Cristina Rovira Gay, Principal Investigator, Predoctoral student, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Vergence VT Protocol
Record Dates: First submitted 2021-11-17; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Vision Disorders; Eye; Movement Disorder (Binocular); Vision Therapy; Binocular Vision Disorder
Keywords: Vergence; Vision Therapy; Binocular Vision
MeSH Terms: conditions — Vision Disorders; Esotropia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Vision Therapy Treatment: vision therapy exercises for fusional vergence abilities (Experimental): The Experimental Group (EG) it consist in a Classical Vision Therapy Treatment. This group will do weekly office-based therapy of 45 minutes of visual exercises during 12 weeks. The office-based done by the EG consists of a vergence therapy and its protocol will follow Scheiman's Protocol and Indications.
  The exercises do not tough the eye or use drugs. They are just visual training exercises that improve fusional convergence and divergence response.
  Interventions: Other: Experimental: Classical Vision Therapy Treatment
- Eye Movement Therapy Treatment: vision therapy placebo exercises not improve fusional vergence (Placebo Comparator): The Control Group or Placebo Group consist in a Control: Eye Movement Therapy Treatment. This group will do weekly office-based placebo therapy of 15 minutes during 12 weeks of visual exercises. This placebo therapy will consist of smooth-pursuit and discrimination exercises that do not influence vergence response.
  The exercises do not tough the eye nor use drugs. They are just visual training exercises that do not improve fusional vergence response as they improve smooth-pursuit eye movements.
  Interventions: Other: Experimental: Classical Vision Therapy Treatment; Other: Control: Eye Movement Therapy Treatment

INTERVENTIONS:
Other: Experimental: Classical Vision Therapy Treatment — Do classical vision therapy treatment for improve vergence
  Other Names: Vision therapy protocol
Other: Control: Eye Movement Therapy Treatment — Do eye movement therapy treatment in order not to improve vergence
  Other Names: Vision therapy protocol
  Arms: Eye Movement Therapy Treatment: vision therapy placebo exercises not improve fusional vergence

SUMMARY:
A vision therapy protocol for vergence ability is mentioned. The purpose of this study is to evaluate objectively the change in the vergence responses of binocular and accommodative normal subjects after performing a classic vision therapy protocol. This study is an interventional, cross-over, and randomized study.

DETAILED DESCRIPTION:
After the first evaluation, subjects will be classified in the Experimental Group (EG) or Control Group (CG) randomly. There will be 18 subjects in each group. A classic vision therapy protocol for fusional vergence will be performed in the EG and the CG will be doing a placebo therapy, based on studies done before.

The EG will do weekly office-based therapy of 45 minutes during 12 weeks and the CG will do weekly office-based placebo therapy of 15 minutes during 12 weeks. This placebo therapy will consist of smooth-pursuit and discrimination exercises that do not influence vergence response. The office-based done by the EG consists of a vergence therapy and its protocol will follow Scheiman's indications protocol. This vision therapy will train both positive and negative fusional vergence amplitudes in the same proportion.

A pre-evaluation, a during evaluation, and a post-evaluation will be done at weeks 1, 6, and 12 respectively to all subjects. After the post-evaluation week, the CG will do 12 weeks more of office-based therapy but, this group will do the same conventional vergence protocol as EG. The CG will be evaluated at week 18, and finally, at week 24.

During the evaluations, the vergence eye movements will be measured during the positive and negative fusional vergence tests. The break and the recovery points will be evaluated to all the subjects with three different methods performed in a randomized order: (1) objective computer-based test in the haploscopic system, (2) prism bar, and (3) phoropter rotary prisms. All these tests will be performed at 40 cm with a classic central visual target.

This study aims to evaluate objectively the change in the vergence responses of binocular and accommodative normal subjects after performing a classic vision therapy protocol.

ELIGIBILITY:
Normal binocular and accommodative subjects will participate in the study. All subjects have to fulfill the inclusion criteria. All evaluations will consist of the following objective and subjective optometric tests, which will be executed for all participants.

1. Monocular and binocular VA at near and distance with their habitual correction
2. Refractive error measured with the Grand Seiko WAM-5500 Autorefractor
3. Cover Test at near (40 cm)
4. Near Point of Accommodation
5. Near Point of Convergence
6. Vergence Facility Test at near (40 cm)
7. Monocular and binocular Accommodation Facility Test at near (40 cm)
8. Negative and Positive Relative Accommodation Test (ARN and ARP)
9. Random Dot 2 Stereo acuity Test
10. CISS questionnaire
11. Fusional Vergence Amplitude using both subjective and objective methods

Exclusion Criteria:

* having eye surgery
* having an eye pathology
* having a binocular or an accommodative disorder
* using orto-K lenses

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-03-29 (Estimated); Study Completion 2022-03-29 (Estimated)

PRIMARY OUTCOMES:
Objective vergence response: To evaluate objectively the change in positive and negative fusional vergence at near of binocularly and accommodative normal subjects after performing a vision therapy | Through study completion, an average of 6 months
  It is measured objectively with an haparoscopic setup and eye movements were recorded with an Eyelink 1000 Plus (SR Research) at 500Hz. Firstly, stimulus disparity changed smoothly at 1PD/s up to 45PD for both divergence (BI) and convergence (BO), mimicking a Risley prism. Secondly, the disparity was changed in steps of 2PD mimicking a prism bar. Break and recovery points were determined offline using a custom Matlab code for the analysis of eye movements.
  Measurements will be compared before and after the therapy treatment.
Subjective vergence response: To evaluate objectively the change in positive and negative fusional vergence at near of binocularly and accommodative normal subjects after performing a vision therapy | Through study completion, an average of 6 months
  It is evaluated with the clinical methods measured subjectively using the Risley prism of the phoropter and the Prism Bar.
  Measurements will be compared before and after the therapy treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Rovira-Gay, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided.

REFERENCES:
- [Result] Scheiman M, Mitchell GL, Cotter S, Cooper J, Kulp M, Rouse M, Borsting E, London R, Wensveen J; Convergence Insufficiency Treatment Trial Study Group. A randomized clinical trial of treatments for convergence insufficiency in children. Arch Ophthalmol. 2005 Jan;123(1):14-24. doi: 10.1001/archopht.123.1.14. PMID 15642806
- [Result] Scheiman M, Talasan H, Alvarez TL. Objective Assessment of Disparity Vergence after Treatment of Symptomatic Convergence Insufficiency in Children. Optom Vis Sci. 2019 Jan;96(1):3-16. doi: 10.1097/OPX.0000000000001320. PMID 30570596
- [Result] Alvarez TL, Scheiman M, Santos EM, Morales C, Yaramothu C, D'Antonio-Bertagnolli JV, Biswal BB, Gohel S, Li X. The Convergence Insufficiency Neuro-mechanism in Adult Population Study (CINAPS) Randomized Clinical Trial: Design, Methods, and Clinical Data. Ophthalmic Epidemiol. 2020 Feb;27(1):52-72. doi: 10.1080/09286586.2019.1679192. Epub 2019 Oct 22. PMID 31640452
- [Result] Scheiman M, Mitchell GL, Cotter S, Kulp MT, Cooper J, Rouse M, Borsting E, London R, Wensveen J. A randomized clinical trial of vision therapy/orthoptics versus pencil pushups for the treatment of convergence insufficiency in young adults. Optom Vis Sci. 2005 Jul;82(7):583-95. doi: 10.1097/01.opx.0000171331.36871.2f. PMID 16044063
- [Result] Scheiman M, Chase C, Borsting E, Mitchell GL, Kulp MT, Cotter SA; CITT-RS Study Group. Effect of treatment of symptomatic convergence insufficiency on reading in children: a pilot study. Clin Exp Optom. 2018 Jul;101(4):585-593. doi: 10.1111/cxo.12682. Epub 2018 Mar 25. PMID 29577409
- [Result] Convergence Insufficiency Treatment Trial Study Group. Randomized clinical trial of treatments for symptomatic convergence insufficiency in children. Arch Ophthalmol. 2008 Oct;126(10):1336-49. doi: 10.1001/archopht.126.10.1336. PMID 18852411